CLINICAL TRIAL: NCT04984356
Title: A Phase 1 Dose-Escalation and Dose-Expansion Study of Anti-CD7 Allogeneic CAR-T Cell Therapy (WU-CART-007) in Patients With Relapsed or Refractory T-cell Acute Lymphoblastic Leukemia (T-ALL)/Lymphoblastic Lymphoma (LBL)
Brief Title: A Phase 1 Study of of Anti-CD7 Allogeneic CAR-T Cell Therapy (WU-CART-007) in Patients With Relapsed or Refractory T-ALL/LBL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wugen, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WU-CART-007 1001; R35CA210084 (NIH); Wugen, Inc. is the sponsor. (Other: Wugen, Inc. is the sponsor.)
Record Dates: First submitted 2021-07-29; First posted 2021-07-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: CAR-T therapy
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: There are two parts to this study, Dose Escalation, and Expansion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- WU-CART-007 (Experimental): A CD7-directed chimeric antigen receptor (CAR) T-cell product.
  A single IV infusion of WU-CART-007 Cells on Day 1 after lymphodepletion
  Interventions: Biological: WU-CART-007

INTERVENTIONS:
Biological: WU-CART-007 — A single IV infusion of WU-CART-007 Cells on Day 1

SUMMARY:
The purpose of this study is to evaluate the safety, recommended dose, and preliminary anti-tumor activity of WU-CART-007 in patients with relapsed or refractory (R/R) T-cell acute lymphoblastic leukemia (T-ALL) or lymphoblastic lymphoma (LBL).

DETAILED DESCRIPTION:
This is a first-in-human, multicenter, Phase 1, single-arm study in patients with R/R T-ALL/T-LBL who have exhausted other treatment options. The study evaluates dose escalation and dose expansion.

ELIGIBILITY:
Key Eligibility Criteria:

* Diagnosed relapsed or refractory T-ALL or T-LBL, as defined by World Health Organization (WHO) classification
* Adequate renal, hepatic, respiratory, and cardiovascular function
* Life expectancy >12 weeks
* ECOG/Karnofsky performance status 0 or 1 at screening (Adults age >16) or Lansky Performance Status 60 and above (adolescents ≤ 16),

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events of WU-CART-007 as assessed by CTCAE v5 | 24 months
  Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of consent until end of study visit
Maximum Tolerated Dose (MTD) | up to 28 days from first dose
  Maximum tolerated or administered dose of WU-CART-007

CONTACTS AND LOCATIONS:
Overall Officials: Cherry Thomas, MD, Study Director — Wugen, Inc.
Locations (12):
- United States (7):
  - City of Hope, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Wisconsin, Madison, Wisconsin
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- France (2):
  - Hospital Saint- Louis, Paris
  - University Hospital Robert Debre, Paris
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - Prinses Maxima Centrum, Utrecht

REFERENCES:
- [Derived] Ghobadi A, Aldoss I, Maude SL, Bhojwani D, Wayne AS, Bajel A, Dholaria B, Faramand R, Mattison RJ, Rijneveld A, Zwaan CM, Calkoen F, Baruchel A, Boissel N, Rettig M, Wood B, Jacobs K, Christ S, Irons H, Capoccia B, Masters D, Gonzalez J, Wu T, Rosario MD, Hamil A, Bakkacha O, Muth J, Ramsey B, McNulty E, Baughman J, Cooper ML, Davidson-Moncada J, DiPersio JF. Phase 1/2 trial of anti-CD7 allogeneic WU-CART-007 for patients with relapsed/refractory T-cell malignancies. Blood. 2025 Sep 4;146(10):1163-1173. doi: 10.1182/blood.2025028387. PMID 40445850
- [Derived] Ghobadi A, Aldoss I, Maude S, Bhojwani D, Wayne A, Bajel A, Dholaria B, Faramand R, Mattison R, Rijneveld A, Zwaan C, Calkoen F, Baruchel A, Boissel N, Rettig M, Wood B, Jacobs K, Christ S, Irons H, Capoccia B, Gonzalez J, Wu T, Del Rosario M, Hamil A, Bakkacha O, Muth J, Ramsey B, McNulty E, Cooper M, Baughman J, Davidson-Moncada J, DiPersio J. Anti-CD7 allogeneic WU-CART-007 in patients with relapsed/refractory T-cell acute lymphoblastic leukemia/lymphoma: a phase 1/2 trial. Res Sq [Preprint]. 2024 Aug 5:rs.3.rs-4676375. doi: 10.21203/rs.3.rs-4676375/v1. PMID 39149468